CLINICAL TRIAL: NCT01706367
Title: A Phase 1, Placebo-Controlled, Randomized, Observer-Blinded Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of A Clostridium Difficile Vaccine Administered With Or Without Adjuvant, In A 3-Dose Regimen In Healthy Adults Aged 50 To 85 Years
Brief Title: Evaluation of a 3-dose Vaccination Regimen With One of Three Ascending Dose Levels of Clostridium Difficile Vaccine With or Without Adjuvant in Healthy Adults Aged 50 to 85 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B5091001
Record Dates: First submitted 2012-09-07; First posted 2012-10-15 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Clostridium Difficile Associated Disease
Keywords: Clostridium difficile; vaccine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Low dose C diff vaccine (Experimental)
  Interventions: Biological: C. difficile vaccine
- Low dose C diff vaccine + adjuvant (Experimental)
  Interventions: Biological: C. difficile vaccine +adjuvant
- Mid dose C diff vaccine (Experimental)
  Interventions: Biological: C. difficile vaccine
- Mid dose C diff vaccine + adjuvant (Experimental)
  Interventions: Biological: C. difficile vaccine +adjuvant
- High dose C diff vaccine (Experimental)
  Interventions: Biological: C. difficile vaccine
- High dose C diff vaccine + adjuvant (Experimental)
  Interventions: Biological: C. difficile vaccine +adjuvant

INTERVENTIONS:
Biological: C. difficile vaccine — 0.5 mL IM injection
  Arms: Low dose C diff vaccine
Biological: C. difficile vaccine +adjuvant — 0.5 mL IM injection
  Arms: Low dose C diff vaccine + adjuvant
Biological: C. difficile vaccine — 0.5 mL IM injection
  Arms: Mid dose C diff vaccine
Biological: C. difficile vaccine +adjuvant — 0.5 mL IM injection
  Arms: Mid dose C diff vaccine + adjuvant
Biological: C. difficile vaccine — 0.5 mL IM injection
  Arms: High dose C diff vaccine
Biological: C. difficile vaccine +adjuvant — 0.5 mL IM injection
  Arms: High dose C diff vaccine + adjuvant

SUMMARY:
This is a first-in-human study (phase 1) of a 3-dose vaccination regimen with one of three dose levels of C difficile vaccine with or without adjuvant in healthy adults aged 50 to 85 years. The main goal of the study is to determine how safe and well-tolerated the vaccine is. In addition, the study aims to assess the immune response to the C difficile vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document.
2. Healthy male and female adults aged 50 to 85 years at enrollment as determined by medical history, physical examination, and the clinical judgment of the investigator to be eligible for the study. Subjects with preexisting chronic medical conditions determined to be stable may be included.
3. Male subjects who, in the opinion of the investigator, are biologically capable of fathering children, and who are sexually active with women of childbearing potential must agree to use a highly effective method of contraception from the time of informed consent through at least 28 days after the last dose of investigational product (through Visit 9 at Month 7).
4. Female subjects who are not of childbearing potential (ie, meet at least one of the following criteria):

   * Have undergone hysterectomy or bilateral oophorectomy;
   * Have medically confirmed ovarian failure or
   * Are medically confirmed to be postmenopausal
5. Availability for the entire duration of the study, and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including completion of the electronic diary (eDiary) from Day 1 to Day 7 following each vaccination.
6. Ability to be contacted by telephone during study participation.

Exclusion Criteria:

1. Previous administration of an investigational C. difficile vaccine or C. difficile monoclonal antibody therapy.
2. Proven or suspected prior episode of CDAD.
3. Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization for worsening disease within 12 weeks before receipt of study vaccine.
4. Serious chronic medical disorders including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) , end stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that in the investigator's opinion precludes the subject from participating in the study.
5. Donation of blood volume of 250 mL or greater, or donation of plasma within 3 months prior to enrollment or during the conduct of the study.
6. Bleeding diathesis or condition associated with prolonged bleeding time that may contraindicate intramuscular injection or blood draw including subjects taking anticoagulant, antiplatelet and/or antithrombotic agents except for low dose daily aspirin (≤325mg per day) within 30 days before enrollment through completion of Visit 9 (Month 7).
7. Any contraindication to vaccination or vaccine components.
8. "Immunocompromised persons or subjects currently on immunosuppressive therapy or with a history of immunosuppressive therapy, including chemotherapy agents for treatment of diseases including, but not limited to cancer, inflammatory bowel disease or autoimmune disease. Recent history (within the past 6 months) of long term (7 days or longer) systemic corticosteroid use."
9. Subjects who received oral or parenteral antibiotics within 1 month before enrollment. Topical antibiotics are allowed.
10. Receipt of blood products or immunoglobulins (including monoclonal antibodies) within 6 months before enrollment through conclusion of the study.
11. Participation in other investigational or interventional studies within 30 days before the current study begins and/or during study participation. Participation in purely observational studies is acceptable.
12. Subjects who are investigational site staff members or relatives of those site staff members, or subjects who are Pfizer employees directly involved in the conduct of the trial.
13. Females of childbearing potential; males of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception for at least 28 days after last dose of investigational product (through Visit 9 at Month 7).
14. Females receiving exogenous estrogen therapy.
15. Residence in a nursing home, long-term care facility, requirement for semiskilled nursing care or assisted living. An ambulatory subject who lives in an autonomous manner in a retirement home or village is eligible for the trial.
16. Any abnormality in screening hematology and/or blood chemistry laboratory values according to the toxicity grading scale. Subjects with stable Grade 1 abnormalities for hemoglobin, leukocyte count, and platelets may be considered eligible at the discretion of the investigator.
17. A positive screening test or known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV).
18. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number subjects reporting local reactions (pain, erythema, and induration) and their severity, as self reported on eDiaries for 7 days following each vaccination. | 7 days
Number of subjects reporting systemic reactions (fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, and new or worsening joint pain) and their severity, as self reported on eDiaries for 7 days following each vaccination. | 7 days
Number of subjects reporting AEs from day 1 (at the time of vaccination) up to 28 days post Dose 3 (visit 9, month 7) and SAEs throughout the study period. | 7 months (AEs) 12 months (SAEs)
Number of subjects with abnormal hematology and blood chemistry laboratory assessments after each vaccination dose. | Day 3, Day 14, Month 1, Day 37, Month 6, Day 187

SECONDARY OUTCOMES:
Neutralizing antibody levels at Month 2. | Month 2
Neutralizing antibody levels after each vaccination dose. | Baseline, Day 14, Month 1, Day 37, Month 6, Day 187, Month 7
Number of subjects in each treatment group with 4 and higher fold-rises in neutralizing antibody levels after each vaccination dose. | Baseline, Day 14, Month 1, Day 37, Month 2, Month 6, Day 187, Month 7
Number of subjects in each treatment group with neutralizing antibody levels ≥ a specified threshold after each vaccination dose. | Baseline, Day 14, Month 1, Day 37, Month 2, Month 6, Day 187, Month 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Cary, North Carolina

REFERENCES:
- [Derived] Sheldon E, Kitchin N, Peng Y, Eiden J, Gruber W, Johnson E, Jansen KU, Pride MW, Pedneault L. A phase 1, placebo-controlled, randomized study of the safety, tolerability, and immunogenicity of a Clostridium difficile vaccine administered with or without aluminum hydroxide in healthy adults. Vaccine. 2016 Apr 19;34(18):2082-91. doi: 10.1016/j.vaccine.2016.03.010. Epub 2016 Mar 15. PMID 26993331
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5091001&StudyName=Evaluation%20of%20a%203-dose%20vaccination%20regimen%20with%20one%20of%20three%20ascending%20dose%20levels%20of%20Clostridium%20difficile%20vaccine%20with%20or%20without%20ad